CLINICAL TRIAL: NCT02356627
Title: The Cancer Home Life Intervention Study Protocol: Effectiveness on Everyday Activities and Quality of Life in People With Advanced Cancer Living at Home. A Randomised, Controlled Multicentre Trial and a Health Economic Evaluation
Brief Title: The Cancer Home Life Intervention Study. A Randomised, Controlled Multicentre Trial and a Health Economic Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Åse Brandt, External lecturer, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AKT
Record Dates: First submitted 2015-01-31; First posted 2015-02-05 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Activities of Daily Living; Everyday Activities; Palliative Care; Cancer; Quality of Life
Keywords: Occupational therapy; Adaptive intervention; Home-based; Assistive Technology; Home modification; Clinical effectiveness; Cost-effectiveness; Cost-utility
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Cancer Home Life Intervention (Experimental): One or more of the following:
  * prioritisation of resources and everyday activities
  * adaptation of activities
  * adaptation of posture and seating positioning
  * provision of assistive devices
  * modification of the physical home environment And usual care from hospital and municipality
  Interventions: Other: The Cancer Home Life Intervention
- Control (No Intervention): Usual care from hospital and municipality

INTERVENTIONS:
Other: The Cancer Home Life Intervention — Adaptive interventions aiming at compensating for functional limitations.
  Arms: The Cancer Home Life Intervention

SUMMARY:
The purpose of this study is to examine the effectiveness and cost-effectiveness of the Cancer Home Life Intervention compared to usual care on performance of and participation in everyday activities and quality of life in people with advanced cancer living at home.

DETAILED DESCRIPTION:
The sample size is based on the primary outcome measure: the mean Activty of Daily Living (ADL) motor ability 1.04 logits (SD 0.727) as measured by the Assessment of Motor and Process Skills (AMPS). A significance level of 0.05 would provide 80% power to detect a between-group difference of 0.3 logits requiring a sample size of N=184. An expected drop-out rate of 32% at 3 months follow-up means that 272 patients with advanced cancer must be included in the study from three hospitals.

Multiple imputation will be used to estimate a plausible value for missing data of participants that are lost to follow-up due to other reasons than death. This does not, however, apply to the primary outcome data where no estimations will be computed.

For normally distributed ratio data the intervention group will be compared with the control group using multiple linear regression analysis of mean changes from baseline. Logistic regression analysis will be used for ordinal data. Adjustments for hospital and for baseline values will be made. A modified intention-to-treat analysis will be applied. Subgroup analyses to identifiy groups that especially benefit from the intervetnion will be performed.

The cost-effectiveness analysis wil be performed with ADL motor ability as the clinical parameter, and the cost-utility analysis will be based on the calculation of Quality Adjusted Life Years (QALY). The Incremental Cost-effectiveness Ratio (ICER) will be calculated and the results summarised in a cost-effectiveness acceptability curve (CEAC).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Diagnosed with cancer
* Evaluated incurable by responsible oncologist in respective out-patient unit
* Functional level 1-2 on the WHO performance scale
* Live within a radius of maximum 60 km from AUH or NH or on the island of Funen
* Live in a private home or in sheltered living
* Know sufficient Danish to fill out questionnaires and participate in interviews.

Exclusion Criteria:

* Cognitive impairment preventing the participants from participating in a structured interview
* Live in a nursing home or a hospice
* Considered incapable of complying with the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Activity of Daily Living (ADL) motor ability as measured by the Assessment of Motor and Process Skills (AMPS) | 3 months
  Observed quality of Activity of Daily Living (ADL) motor ability

SECONDARY OUTCOMES:
Individually Prioritised Problems Assessment (IPPA) | 6 weeks and 3 months
  Everyday activities that the participant has problems with and prioritise to have solved
Everyday activity pattern captured by a One Day Diary | 3 months
  The participant records every ½ hour what he/she does, where, is together with, how he/she feels mentally and physically
Impact on Participation and Autonomy Questionnaire (IPAQ) | 6 weeks and 3 months
  Autonomy and participation is assessed regarding autonomy indoors, family roles, and social life and relationships
The European Organization for Research Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ C-30) | 6 weeks and 3 months
  Cancer specific health-related quality of life
EuroQol 5-dimensions 5 levels (EQ-5D-5L) | 6 weeks, 3 months, and 6 months
  Health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Karen la Cour, PhD, Principal Investigator — University of Southern Denmark; Åse Brandt, PhD, Principal Investigator — The National Bord of Social Services
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandt Å, la Cour K, Wæhrens. Activity problems important to people with advanced cancer living at home. Oral session presented at: 16th International Congress of the World Federation of Occupational Therapists.; June 18-21; Yokohama, Japan; 2014.
- [Background] Johnsen AT, Petersen MA, Pedersen L, Houmann LJ, Groenvold M. Do advanced cancer patients in Denmark receive the help they need? A nationally representative survey of the need related to 12 frequent symptoms/problems. Psychooncology. 2013 Aug;22(8):1724-30. doi: 10.1002/pon.3204. Epub 2012 Oct 8. PMID 23042603
- [Background] la Cour K, Johannessen H, Josephsson S. Activity and meaning making in the everyday lives of people with advanced cancer. Palliat Support Care. 2009 Dec;7(4):469-79. doi: 10.1017/S1478951509990472. PMID 19939309
- [Background] la Cour K, Nordell K, Josephsson S. Everyday lives of people with advanced cancer: Activity, time, location, and experience. OTJR Occup Part Health 2009 December;29(4):154-162.
- [Background] Lindahl-Jacobsen L. Occupational therapy for cancer patients - a randomised, controlled study [PhD thesis]. Research Unit of General Practice, Institute of Public Health: University of Southern Denmark; 2014.
- [Background] Rabow M, Kvale E, Barbour L, Cassel JB, Cohen S, Jackson V, Luhrs C, Nguyen V, Rinaldi S, Stevens D, Spragens L, Weissman D. Moving upstream: a review of the evidence of the impact of outpatient palliative care. J Palliat Med. 2013 Dec;16(12):1540-9. doi: 10.1089/jpm.2013.0153. Epub 2013 Nov 13. PMID 24225013
- [Background] Sviden GA, Tham K, Borell L. Involvement in everyday life for people with a life threatening illness. Palliat Support Care. 2010 Sep;8(3):345-52. doi: 10.1017/S1478951510000143. PMID 20875178
- [Background] Vendrusculo Fangel LM, Sanches Panobianco M, Martins Kebbe L, de Almeida AM, de OG. Qualify of life and daily activities performance after breast cancer treatment. ACTA PAUL ENFERMAGEM 2013 February;26(1):93-100.
- [Background] Wæhrens E, la Cour K, Brandt Å. The quality of ADL task performance based on self-report and observation in people living at home with cancer. Poster presented at: 16th International Congress of the World Federation of Occupational Therapists.; June 18-21; Yokohama, Japan; 2014.
- [Derived] Oestergaard LG, la Cour K, Lindahl-Jacobsen LE, Brandt A, Pilegaard MS. The Cost-Effectiveness of the Cancer Home-Life Intervention: An Economic Evaluation Alongside a Randomized Clinical Trial with a Six-Month Time Frame. J Palliat Med. 2025 Dec;28(12):1620-1628. doi: 10.1177/10966218251374527. Epub 2025 Sep 16. PMID 40955537
- [Derived] la Cour K, Gregersen Oestergaard L, Brandt A, Offersen SMH, Lindahl-Jacobsen L, Cutchin M, Pilegaard MS. Process evaluation of the Cancer Home-Life Intervention: What can we learn from it for future intervention studies? Palliat Med. 2020 Dec;34(10):1425-1435. doi: 10.1177/0269216320939227. Epub 2020 Jul 2. PMID 32611224
- [Derived] Pilegaard MS, la Cour K, Gregersen Oestergaard L, Johnsen AT, Lindahl-Jacobsen L, Hojris I, Brandt A. The 'Cancer Home-Life Intervention': A randomised controlled trial evaluating the efficacy of an occupational therapy-based intervention in people with advanced cancer. Palliat Med. 2018 Apr;32(4):744-756. doi: 10.1177/0269216317747199. Epub 2018 Jan 4. PMID 29299957
- [Derived] Brandt A, Pilegaard MS, Oestergaard LG, Lindahl-Jacobsen L, Sorensen J, Johnsen AT, la Cour K. Effectiveness of the "Cancer Home-Life Intervention" on everyday activities and quality of life in people with advanced cancer living at home: a randomised controlled trial and an economic evaluation. BMC Palliat Care. 2016 Jan 22;15:10. doi: 10.1186/s12904-016-0084-9. PMID 26801394